CLINICAL TRIAL: NCT00886743
Title: Study Of The Effects Of Oprelvekin On Cardiac Repolarization In Subjects At Risk Of Severe Thrombocytopenia After Myelosuppressive Chemotherapy
Brief Title: Study Evaluating The Effects Of Oprelvekin On Cardiac Repolarization In Subjects With Chemotherapy Induced Thrombocytopenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reason, Pfizer's requested withdrawal of the Biologics License Application (BLA) . This study is not being discontinued for efficacy or safety reason
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3067K1-2213; B2491001 (Other: Alias Study Number)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Severe Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — oprelvekin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oprelvekin as subcutaneous injection (50 mg/kg once daily) (Other): Open label treatment with oprelvekin
  Interventions: Drug: oprelvekin

INTERVENTIONS:
Drug: oprelvekin — injection, 50 mg/kg, once daily

SUMMARY:
This is an open-label study in which oprelvekin will be administered for the prevention of severe low blood platelet cell counts (cells in your blood that keep bleeding and clotting stable) in adults with cancer who are taking chemotherapy (anti-cancer drug) that has a side effect of blocking your bone marrow from making platelet cells. The purpose of this study is to learn more about the effects of the recommended dose of oprelvekin on the heart's electrical cycle.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be 18 to 65 years of age, with nonmyeloid malignancies for whom oprelvekin is indicated.
* At least one documented occasion of adequate hematologic recovery from previous or current chemotherapy.
* Adequate renal and hepatic excretory function.

Exclusion Criteria:

* A marked baseline prolongation of QT/QTc interval (eg, repeated [two out of three readings] demonstration of a QTcF interval >450 msec.
* Additional risk factors for torsades de pointes including heart failure (subjects that have functional class III or IV congestive heart failure), hypokalemia, hypomagnesemia, or hypocalcemia.
* A pace maker or defibrillator.
* A history of LQTS, syncope, seizure, or the unexplained cardiac-related death of a family member at less than 30 years of age.
* Requirement of concomitant prescription or non-prescription medications or dietary supplements that have a risk of causing torsades de pointes or prolonged QT/QTc interval.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - Pfizer Investigational Site, Santa Monica, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Howard University, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Gabrail Cancer Center Research, Canton, Ohio
  - Pfizer Investigational Site, Canton, Ohio
  - Gabrail Cancer Center Research, Dover, Ohio
  - Pfizer Investigational Site, Dover, Ohio
  - Pfizer Investigational Site, Middletown, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Pfizer Investigational Site, Laredo, Texas
  - South Texas Research Alliance LLC., Laredo, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3067K1-2213&StudyName=Study%20Evaluating%20The%20Effects%20Of%20Oprelvekin%20On%20Cardiac%20Repolarization%20In%20Subjects%20With%20Chemotherapy%20Induced%20Thrombocytopenia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants were screened; of these, 19 received treatment.
Groups:
- Oprelvekin, 50 μg/kg: Participants received 50 μg/kg of oprelvekin once daily by subcutaneous injection.
Period: Overall Study
Arm/Group | Oprelvekin, 50 μg/kg
Started | 19 (Received treatment)
Completed | 15
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: All participants who had received at least 1 dose of oprelvekin.
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 17
  Black or African American | 2
Weight [Mean (Standard Deviation); unit: Kilograms] | 76.9 (25.7)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms/meters^2] | 26.7 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Time-matched Change From Baseline in Corrected QT Interval Using a Population-specific Correction Formula (QTcN)
Description: Because the sponsor terminated the study prematurely, this population-specific correction of QT was not done. QT data collected during the study corrected using the Bazett's and Fridericia formulae are presented as secondary outcome measures.
Time Frame: Postdose Day 1 to end of treatment
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Time-matched Change From Baseline in Corrected QT (QTc) Interval ≥30 or 60 Msec Using Fridericia's (QTcF) and Bazett's (QTcB) Correction Formulas
Description: Based on average across triplicates for a given hourly measurement.
Time Frame: Postdose Day 1 to end of treatment
Population: Participants who completed baseline and postdose triplicate electrocardiograms through at least 3 continuous days of dosing. Those who received any systemic concomitant medications that had the potential for drug interaction and sporadic effect on QT/QTc data, and thus impacted results, were excluded from the analyses.
Measure: Number; unit: Participants
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 19
Participants
  QTcF change ≥30 msec | 5
  QTcF change ≥60 msec | 0
  QTcB change ≥30 msec | 9
  QTcB change ≥60 msec | 2

3. Secondary Outcome: Number of Participants With Corrected QT (QTc) Interval ≥450, ≥480, and ≥500 Msec Using Bazett's (QTcB) and Fridericia's (QTcF) Correction Formulas
Description: Definition of QTc is based on observed individual values rather than the average across triplicate starting from Day 1 postdose through the end of treatment.
Time Frame: Postdose Day 1 to end of treatment
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 19
Participants
  QTcF ≥450 msec | 2
  QTcF ≥480 msec | 0
  QTcF ≥500 mec | 0
  QTcB ≥450 msec | 13
  QTcB ≥480 msec | 3
  QTcB ≥500 mec | 1

4. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Oprelvekin
Description: Cmax was obtained directly from the serum oprelvekin concentration data using noncompartmental methods.
Time Frame: Postdose Day 1 to end of treatment
Population: All participants who received at least 1 dose of study drug and had at least 1 concentration assessment.
Measure: Number; unit: picograms/mililiter
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 11
picograms/mililiter
  Participant 1 | 15900
  Participant 2 | 20100
  Participant 3 | 20200
  Participant 4 | 17000
  Participant 5 | 12200
  Participant 6 | 19100
  Participant 7 | 17300
  Participant 8 | 17500
  Participant 9 | 34500
  Participant 10 | 25000
  Participant 11 | 24000

5. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Oprelvekin
Description: Tmax was obtained directly from the serum oprelvekin concentration data using noncompartmental methods.
Time Frame: Postdose Day 1 to end of treatment
Population: All participants who received at least 1 dose of study drug and had at least 1 concentration assessment.
Measure: Number; unit: hours
Arm/Group | Oprelvekin, 50 μg/kg
Number analyzed (Participants) | 11
hours
  Participant 1 | 1
  Participant 2 | 4
  Participant 3 | 6
  Participant 4 | 3
  Participant 5 | 5
  Participant 6 | 3
  Participant 7 | 3
  Participant 8 | 6
  Participant 9 | 3
  Participant 10 | 3
  Participant 11 | 2

ADVERSE EVENTS:
Arm/Group | Oprelvekin, 50 μg/kg
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oprelvekin, 50 μg/kg (N=19)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oprelvekin, 50 μg/kg (N=19)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
QRS axis abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Short QT Interval with ST changes (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.